CLINICAL TRIAL: NCT00095719
Title: A Safety & Tolerability Study of Intramuscular Aripiprazole in Acutely Agitated Patients Diagnosed With Dementia
Brief Title: Intramuscular Aripiprazole in Acutely Agitated Patients Diagnosed With Dementia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN138-131
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2008-08

CONDITIONS: Dementia; Alzheimer's Disease
Keywords: Acute agitation in patients diagnosed with Dementia
MeSH Terms: conditions — Dementia; Alzheimer Disease | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A1 (Active Comparator)
  Interventions: Drug: Aripiprazole
- B1 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aripiprazole — IM Solution, IM, Cohort 1 - 2.5mg (.33cc) maximum dose 5.0mg; 2 injections 2nd injection 2 hours after first; Cohort 2 - 5.0mg (.67cc) maximum dose 10 mg; 2 injections 2nd injection 2 hours after first; Cohort 3 - 10 mg (1.3cc) or 5.0 mg (.67cc) maximum dose 15mg; 1 injection, 24 hour observation for all cohorts.
  Other Names: Abilify
  Arms: A1
Drug: Placebo — IM Solution, IM, Cohort 1 - 0mg; 2 injections 2nd injection 2 hours after first; Cohort 2 - 0mg; 2 injections 2nd injection 2 hours after first; Cohort 3 - 0mg; 1 injection, 24 hour observation for all cohorts.
  Arms: B1

SUMMARY:
The purpose of this trial is to test the safety & tolerability of intramuscular aripiprazole in acutely agitated patients diagnosed with Dementia.

ELIGIBILITY:
Inclusion Criteria:

* Acute agitation in Patients with a DSM-IV diagnosis of Alzheimer's, vascular or mixed Dementia.

Exclusion Criteria:

* Current DSM-IV Axis 1 diagnosis other than Alzheimer's, vascular or mixed Dementia.

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125
Dates: Start 2003-12; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
tolerability

SECONDARY OUTCOMES:
safety assessments

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (14):
- United States (14):
  - Local Institution, Santa Ana, California
  - Local Institution, Hamden, Connecticut
  - Local Institution, Hialeah, Florida
  - Local Institution, Miami, Florida
  - Local Institution, North Miami, Florida
  - Local Institution, Indianapolis, Indiana
  - Local Institution, New York, New York
  - Local Institution, Staten Island, New York
  - Local Institution, Dayton, Ohio
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Tulsa, Oklahoma
  - Local Institution, Hershey, Pennsylvania
  - Local Institution, Austin, Texas
  - Local Institution, Midvale, Utah